CLINICAL TRIAL: NCT02870075
Title: The Influence of Different Dietary Status on the Acute Responses to Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bath (Other)
Collaborators: Ministry of Education, Taiwan (Other Government)
Responsible Party: Principal Investigator, Yung-Chih Chen, PhD student, University of Bath
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 13/SW/0020
Record Dates: First submitted 2016-02-09; First posted 2016-08-17 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Adipose Tissue Gene Expression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fed exercise (Active Comparator): Fed prior to exercise
  Interventions: Behavioral: Fed exercise
- Fasted exercise (Active Comparator): Fasted prior to exercise
  Interventions: Behavioral: Fasted exercise

INTERVENTIONS:
Behavioral: Fed exercise — Participants consumed a meal (Fed) 2 h prior to 1 h moderate intensity exercise at 60% VO2max.
  Arms: Fed exercise
Behavioral: Fasted exercise — Participants remained fasting (Fasted) 2 h prior to 1 h moderate intensity exercise at 60% VO2max.
  Arms: Fasted exercise

SUMMARY:
The purpose of this study is to investigate whether dietary conditions (fed versus fasted) affects the acute responses to exercise.

DETAILED DESCRIPTION:
Pre-trial assessments

V̇O2max measurement V̇O2max was determined using an incremental continuous treadmill test until the point of volitional exhaustion. For most participants, a treadmill speed of 4 km/h and gradient of 8.5% was chosen. Participants were tested at this speed and gradient with the speed increased by 1 km/h after every 3 min stage. One minute expired air samples were collected into Douglas bags (Douglas Bags, Hans Rudolph, MO, USA), and RPE and heart rates were measured in the final minute of each stage and also at the point of volitional exhaustion, defined as when the participant indicated that only 1 min remained until fatigue. Samples were analysed for relative expired fractions of oxygen and carbon dioxide gas (Servomex, Crowborough, UK) and the total volume with in the bag was measured using a dry gas meter (Harvard Apparatus, Kent, UK).

Physical activity assessment Participants wore a combined heart rate/accelerometer monitor for one week to assess their habitual physical activity energy expenditure (Actiheart, Cambridge Neurotechnology Ltd., Cambridge, UK). This was attached to the left chest via 2 adhesive ECG pads for 24 hours per day except for during showering/bathing/swimming.

Body composition analysis Body mass was measured using digital scales post-void (TANITA corp., Tokyo, Japan). Waist and hip circumference was assessed according to World Health Organisation guidelines. Body composition was determined using Dual energy X-ray absorptiometry (Discovery, Hologic, Bedford, UK). Abdominal subcutaneous and visceral adipose tissue mas was estimated from a central region between L1-L4.

Trial days In the 72 h prior to each main trial, participants were asked to refrain from performing any strenuous physical activity and from consuming alcohol/caffeine for 48 h prior to the main trials. A dietary record was completed 48 h before the first main trial and participants were asked to replicate this diet prior to their second main trial.

On main trial days, participants arrived at the laboratory between 8-9am following a 12 h fast. After anthropometric measurements, participants rested on a bed for 15 minutes, followed by four 5 min expired gas samples collections to determine resting metabolic rate (RMR) using substrate oxidation under resting conditions.

Participants then either consumed a meal (FED) or remained fasting (FASTED) and cannula blood samples were taken every 15 minutes for the following 60 minutes. A further blood sample was collected at 120 min immediately before the walking protocol. In both the FASTED and FED treatments, participants walked on the treadmill at 60% V̇O2max for 60 minutes and one minute of expired air samples, ratings of perceived exertion (RPE) and heart rate were collected at 5, 20, 40 and 60 minutes. After finishing the exercise, another blood sample was immediately collected and participants then rested for a further 60 minutes. At this point, a second adipose tissue and final blood sample was taken.

Adipose tissue culture and gene expression After adipose tissue biopsy and cleaning, tissue was minced to approximately 5-10 mg and directly placed in sterile culture plates (Nunc, Roskilde, Denmark) with endothelial cell basal media (ECBM) containing 0.1% fatty acid-free bovine serum albumin 100 U ml-1 penicillin and 0.1 mg ml-1 streptomycin (Sigma-Aldrich, Gillingham, UK). Adipose tissue was incubated with a final ratio of 100mg tissue per 1 ml ECBM media for 3 hours. A 37°C, 5% CO2 and 95 ± 5% relative humidity incubator was used (MCO-18A1C CO2 incubator; Sanyo, Osaka, Japan). Media was transferred to sterile eppendorfs and stored at -80°C after 3 hours incubation. Approximately 200 mg adipose tissue was homogenised in 5ml Trizol in an RNase/DNase-free sterile tube (Invitrogen, Paisley, UK) and stored at -80°C before further analysis.

Sample size There is no data regarding how different dietary status (fed versus fasted) affects the acute responses to exercise on overweight males. However, a previous study using a similar meal showed that feeding had an enormous effect on the use of lipid during exercise - and thus indicates that the role of adipose tissue during exercise would be potentially very different. In order to see an effect on lipid oxidation during exercise with 95% power and 5% alpha, we would require 6-8 participants. To ensure that these results are generalizable and also to account for greater variability in other outcome, we recruited a total 10 participants from the study.

Statistics:

All data was presented as mean ± standard error of mean (SEM). Incremental area under curve (iAUC) was calculated using the trapezoid method and differences between trials analysed using paired t-tests. Glucose, insulin, NEFA, TAG, adipokines, and cell culture outcomes were determined using a two-way ANOVA with repeated measures using SPSS version 22 (IBM, Armonk, NY, USA). Where significant interactions (trial × time) were found, a post hoc analysis was applied using t-test with the Holm-Bonferroni correction. Single comparisons used a t-test or non-parametric equivalent. Statistical significance was set at p ≤ 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Aged between 18 to 35 years
* Central overweight (waist circumference 94-128 cm)
* Weight stable for more than 3 months (no change in weight +/- 3%)
* Non-smoker
* Able to walk for a long period of time

Exclusion Criteria:

* Personal history of/existing diabetes, cardiovascular disease, metabolic disease or dyslipidaemia
* Waist circumference < 94cm and >128cm
* Taking medications that may influence lipid or carbohydrate metabolism or immune system function
* Unable to take part in structured exercise for any reason (e.g., injury or disability) or a positive response to any questions on the Physical Activity Readiness questionnaire (PAR-Q)

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2013-05; Primary Completion 2014-10 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Changes in gene expression in the adipose tissue | Before the meal and 1 h after exercise (255 minutes)

SECONDARY OUTCOMES:
Changes in insulin, glucose, TAG and NEFA in blood | 255 minutes
Changes in serum Interleukin-6 (IL-6), leptin and adiponectin | 255 minutes
Changes in Interleukin-6 (IL-6), leptin and adiponectin protein secretion from adipose tissue explants | Before the meal and 1 h after exercise (255 minutes)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chen YC, Travers RL, Walhin JP, Gonzalez JT, Koumanov F, Betts JA, Thompson D. Feeding influences adipose tissue responses to exercise in overweight men. Am J Physiol Endocrinol Metab. 2017 Jul 1;313(1):E84-E93. doi: 10.1152/ajpendo.00006.2017. Epub 2017 Mar 14. PMID 28292758